CLINICAL TRIAL: NCT04584541
Title: Study of the Viral Load and Humoral and Cellular B and T Responses in Patients With Rheumatoid Arthritis and Spondyloarthritis Under Immunosuppressive Treatments
Brief Title: SarS-Cov-2 Viral Infection (COVID-19) in Patients With Chronic Inflammatory Rheumatism
Acronym: COVIRIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study of the long term antibody response is no longer relative due to the introduction of Covid vaccine.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200598
Record Dates: First submitted 2020-06-10; First posted 2020-10-14 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Spondyloarthritis; Rheumatoid Arthritis; Covid19
Keywords: Spondyloarthritis; Rheumatoid arthritis; Immunosuppressive treatments; COVID19; Sars-Cov-2
MeSH Terms: conditions — Spondylarthritis; Arthritis, Rheumatoid; COVID-19 | interventions — Hematologic Tests; Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Other): Index cases (RA and SpA patients under immunosuppressive treatments)
  Interventions: Biological: blood tests; Biological: Nasopharyngeal swabs; Biological: Stools
- controls (Other): Members of index cases family cluster infected with the same viral strain
  Interventions: Biological: blood tests; Biological: Nasopharyngeal swabs; Biological: Stools

INTERVENTIONS:
Biological: blood tests — Memory T and B cell response assessment Humoral response assessment (Specific anti-Sars-Cov-2 antibodies characterization)
  Other Names: Immune response assessment
Biological: Nasopharyngeal swabs — SarS-Cov-2 viral load assessment
Biological: Stools — SarS-Cov-2 viral load assessment

SUMMARY:
The purpose of this study is to assess whether immunosuppressive therapies used by patients with chronic inflammatory rheumatic diseases have an impact on the viral load and the humoral and cellular responses during viral infection with SarSCoV2, compared to members of their family cluster infected with the same viral strain.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) and spondyloarthritis (SPA) are the two most common chronic inflammatory rheumatic diseases, with a prevalence of 0.5-1% for RA and about 0.35% for SPA. Many studies have described an increased risk of serious infectious diseases directly associated with increased morbidity and mortality among those patients. This increased risk (frequency and severity) results from the disease itself, especially if the rheumatism is not controlled with high disease activity, but also due to the immunosuppressive treatments used to treat these patients. The risk of infection is measured by the Incidence Rate (IR) corresponding to the number of events (infections) per 100 patients/years of follow-up. This risk is accepted as comparable between patients with SpA or RA and ranges from 22 to 34/100 patient-years, depending on the studies, for patients on biologics. The risk of infection is higher for patients on biotherapy than for patients on Disease Modifying Anti-Rheumatic Drugs (DMARDs - mainly Methotrexate) and the combination of corticosteroid therapy with the biotherapies further increases this risk of infection. Lung and upper respiratory tract infections are the most common infections observed under biotherapy. The risk of infection may be different depending on the biotherapy considered. Moreover, the vaccine response is also highly variable depending on the biotherapy, treatments with Rituximab, methotrexate and abatacept being those interfering the most with the quality of the vaccine response. The working hypothesis is therefore that certain immunosuppressive treatments used in these inflammatory rheumatic conditions may interfere with the humoral and/or cellular anti-SarS-Cov-2 immune response.

Since December 2019, the first SARS-Cov-2 (Severe acute respiratory coronavirus 2 syndrome) infections have been described in Wuhan province in China. In April 2020, 1,824,950 people were officially infected in 193 countries worldwide with 112,510 deaths reported (Agence France Presse and World Health Organization; 13 April 2020). To date, the investigators have a limited amount of data concerning the seroconversion of infected subjects, the protective or non-protective nature of the specific antibodies generated, and the duration of protection. No data have been generated on the specific B and T responses of SarS-Cov-2. In addition, the few available data in the literature on SarS-Cov-2 only concern the general population, not exposed to immunosuppressive treatments.

However, major questions are currently unanswered for patients on immunosuppressive treatments: Are they excreting the virus for longer periods of time? How long can this viral excretion be measured in the upper airways and in the stool? Do they develop a humoral and cellular immune response similar to the general population? Accurate knowledge of the dynamics of the virus and the immune response induced will be essential for the development of strategies for antiviral treatment, vaccination protocols and for the epidemiological control of Covid-19.

ELIGIBILITY:
Inclusion Criteria:

cases

* Patient with spondyloarthritis fulfilling the ASAS criteria
* Patients with rheumatoid arthritis fulfilling the ACR/EULAR criteria and
* Immunosuppressive therapy: Methotrexate, leflunomide, anti-TNF, Anti-IL6R, abatacept, rituximab, Jak inhibitors (tofacitinib or baricitinib) And
* infected with the SarS-Cov-2 (positive PCR and/or serology and/or CT-scan)

Controls:

* Family cluster member confined to the same location as the index subject
* Infected with the SarS-Cov-2 (positive PCR and/or serology and/or CT-scan)

Exclusion Criteria:

cases and controls

* Pregnant woman
* Breastfeeding woman
* Immunosuppressed subject for members of the familiar cluster of the index subject
* Patient with no social security
* Patients whose freedom is limited by the judicial or administrative authority
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Detection of SarS-Cov-2 RNA in feces and nasopharyngeal swabs | up to Day 30
  Nasopharyngeal swabs : Detection of SarS-Cov-2 RNA
Detection of SarS-Cov-2 RNA in feces and nasopharyngeal swabs | between Day 30 and Day 90
  Nasopharyngeal swabs : Detection of SarS-Cov-2 RNA
Detection and quantification of IgG, IgM and IgA specific for SarS-Cov-2 N and S proteins in blood | up to Day 30
Detection and quantification of IgG, IgM and IgA specific for SarS-Cov-2 N and S proteins in blood | between Day 30 and Day 90
Detection and quantification of IgG, IgM and IgA specific for SarS-Cov-2 N and S proteins in blood | 6 Months
Detection and quantification of IgG, IgM and IgA specific for SarS-Cov-2 N and S proteins in blood | 12 Months
Detection and quantification of IgG, IgM and IgA specific for SarS-Cov-2 N and S proteins in blood | 24 Months
Isolation and characterization of B and T lymphocytes in blood | up to Day 30
Isolation and characterization of B and T lymphocytes in blood | between Day 30 and Day 90
Isolation and characterization of B and T lymphocytes in blood | 6 Months
Isolation and characterization of B and T lymphocytes in blood | 12 Months
Isolation and characterization of B and T lymphocytes in blood | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Miceli-Richard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No